CLINICAL TRIAL: NCT01001936
Title: Phase 1 Does-escalation Study of Oral SKI-606 in Subjects With Advanced Malignant Solid Tumors
Brief Title: Study Evaluating SKI-606 in Subject With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3160A1-102
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2009-10-27 (Estimated); Status verified 2009-10

CONDITIONS: Tumors
Keywords: PHASE 1 SKI-606 Solid tumor
MeSH Terms: conditions — Neoplasms | interventions — bosutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: SKI-606

INTERVENTIONS:
Drug: SKI-606

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of oral SKI-606 (100, 200, 300 or 400 mg) administered on a daily schedule to subjects with advanced malignant solid tumors and to define a maximum tolerated dose (MTD) in this subject population. This study will also obtain preliminary information on the pharmacokinetics and antitumor activity of orally administered SKI-606 in subjects with advanced malignant solid tumors

ELIGIBILITY:
Inclusion Criteria:

1. Advanced or recurrent solid malignancy confirmed histologically or cytologically for which no effective therapy is available
2. Recovery from acute adverse effects of prior therapies to £ Grade 1 (excluding alopecia)
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 - 1
4. Adequate hepatic, renal, and bone marrow function
5. Age 20 to 74 years
6. Willingness of male and female subjects, who are not surgically sterile or postmenopausal, to use reliable methods of birth control for the duration of the study and for 6 months and 30 days after the last dose of test article for male and female, respectively
7. Life expectancy of at least 12 weeks

Exclusion Criteria:

1. Use of any systemic antitumor agents or any investigational agent within 28 days before the enrollment (42 days if the previous chemotherapy included nitrosoureas or mitomycin C)
2. Ongoing clinical requirement for administration of a strong inhibitor of CYP3A4
3. Prior exposure to SKI-606 or any other Src-kinase inhibitor
4. Major surgery or radiotherapy within 2 weeks before the enrollment (recovery from previous surgery should be complete before day 1)
5. Subjects unable or unwilling to swallow SKI-606 capsules
6. Active central nervous system (CNS) metastases, as indicated by clinical symptoms, cerebral edema, requirement for corticosteroids and/or progressive growth
7. Recent or ongoing clinically-significant gastrointestinal disorder
8. Pregnant or breastfeeding women
9. Subjects who meet the following criteria:

   * Evidence of serious active infection, significant medical or psychiatric illness
   * History of unexplained syncope or known ventricular arrythmia
   * Known seropositivity to HIV, or current or chronic Hepatitis B or Hepatitis hepatitis C
   * Hypokalemia
   * Unstable concurrent medical conditions
   * Any other condition that, in the investigator's judgment, make the subject inappropriate for this study the subject inappropriate for this study

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Safety as measured by AE information. Tolerability as measured by DLT observation. | 2 years

SECONDARY OUTCOMES:
Pharmacokinetics as measured by Taylor Technology Antitumor activity as measured by RECIST | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer